CLINICAL TRIAL: NCT04851912
Title: Preclinical Development of a Speech-based Digital Biomarker for Psychiatric Disease
Brief Title: Speech-based Digital Biomarker for Psychiatric Disease
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Winterlight Labs (Industry)
Responsible Party: Sponsor
Other Study IDs: WLL-PRO-005
Record Dates: First submitted 2021-04-12; First posted 2021-04-21 (Actual); Last update posted 2022-09-27 (Actual); Status verified 2022-09

CONDITIONS: Speech; Psychiatric Disorder; Language
MeSH Terms: conditions — Speech; Mental Disorders; Language

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- General: Participants with or without psychiatric disorders
  Interventions: Other: Winterlight Apps

INTERVENTIONS:
Other: Winterlight Apps — Longitudinal speech recordings

SUMMARY:
The general objectives of this study are to build a proof-of-concept, speech-based, digital biomarker for identifying the presence and tracking the severity of psychiatric disease.

DETAILED DESCRIPTION:
The purpose of this study is to gather longitudinal data to examine how speech features and symptoms change over different intervals of time and the reliability of repeated, high frequency test administration. Participants will complete a variety of speech and language tasks using the Winterlight Assessment (iOS app) everyday for 30 days. The following is the list of assessments that participants will complete; 1) Daily assessment of mood, 2) Winterlight assessment which contains a series of verbal response tasks where participants are recorded through a tablet app, and 3) Clinical assessments.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female adults aged 18 to 95.
* English as a first language, or English as a second language with conversational proficiency.
* Own an iOS device (iPhone or iPad) and willing to install the study app.
* A reliable (cellular or WiFi) home internet connection and accessible email address

Exclusion Criteria:

* Residence outside of Canada or the United States.
* Clinically significant vision impairment (corrected vision is acceptable).
* Clinically significant hearing impairment (use of hearing aids is acceptable)

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Anyone who does not have hearing or vision impairment.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-04-27 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Speech recordings | Everyday for 30 business days until study completion, about 2 years
  500+ features to be extracted from each recording

SECONDARY OUTCOMES:
Depression scores | Everyday for 30 business days until study completion, about 2 years
  Depression and depression like scores to be collected through surveys

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Robin, PhD, Principal Investigator — Clinical Research Director, Winterlight Labs
Locations (1):
- Winterlight Labs, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided